CLINICAL TRIAL: NCT07360626
Title: Effectiveness of an Exercise and Health Education Program for Health Promotion in Textile Workers: A Pre-Post Intervention Study
Brief Title: Exercise and Health Education for Textile Workers: A Pre-Post Study
Acronym: LACOR-HEALTH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7/1/25-26
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Musculoskeletal Disorders (MSDs); Musculoskeletal Diseases or Conditions
Keywords: Textile workers; Exercise program; Health education; Pre-post intervention
MeSH Terms: conditions — Musculoskeletal Diseases; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Exercise and Health Education Program (Experimental): Participants in this arm will receive an eight-week physical therapy and health education program. Exercise sessions will be held twice weekly for 20 minutes via the RehBody mobile app, focusing on mobility, strength, and stability of the upper and lower extremities. Participants will also attend weekly 45-minute in-person workshops covering pain management, coping strategies, self-efficacy, stress management, relaxation, sleep hygiene, and healthy habits.
  Interventions: Other: Combined Exercise Training and Health Education Program

INTERVENTIONS:
Other: Combined Exercise Training and Health Education Program — The intervention consists of an 8-week hybrid program combining exercise training and workplace-based health education. Eight on-site educational workshops (one per week) are delivered during working hours and address topics related to pain management, physical activity, stress management, and healthy lifestyle behaviors, including review and discussion sessions.
  The exercise training includes two weekly sessions delivered through a mobile application (RehBody platform). Sessions begin with a warm-up incorporating mobility and core exercises, followed by strengthening exercises for the upper and lower extremities. Exercise difficulty progresses from bilateral, single-joint movements to unilateral, multi-joint exercises. The program is delivered by trained physical therapists and is adaptable to individual participant needs.

SUMMARY:
Musculoskeletal disorders (MSDs) significantly impact quality of life, health status, and work ability. Standard treatments include ergonomic interventions, therapeutic exercise programs, education on risk prevention, active breaks, and physiotherapy. This study aims to assess the current physical and psychosocial condition of textile manufacturing workers and to evaluate the impact of a combine exercise and health education program on their physical and psychosocial outcomes.

The eight-week intervention consists of a weekly in-person workshops and two asynchronous online exercise sessions per week via a mobile app, with exercises adjusted based on participant feedback.

Participants will be recruited from voluntary textile workers at Lacor Textil, S.L., aged 18-65, with active employment. All participants will receive the intervention program.

Primary objectives are to assess the baseline physical and psychosocial condition of participants and to evaluate the effects of the eight-week intervention on their physical fitness, musculoskeletal health, and overall psychosocial well-being

Secondary objectives are to examine changes in the intensity and location of musculoskeletal pain and discomfort, the prevalence of symptoms in different body regions, upper and lower body strength using standardized tests, work ability and perception of work performance, and psychosocial and cognitive factors including sleep quality, stress, anxiety, depression, productivity, and quality of life.

Hypothesis: The implementation of an eight-week physical exercise and health education program in textile workers will reduce perceived musculoskeletal discomfort and pain, and improve their physical fitness and psychosocial well-being.

DETAILED DESCRIPTION:
The protocol uses a quasi-experimental, single-group pre-post design without a control group, conducted in a real occupational setting. All participants will undergo an 8-week intervention program, followed by a 4-week follow-up period. The intervention adopts a hybrid format, combining face-to-face sessions at the workplace with asynchronous online exercise sessions delivered through a mobile application.

Prior to the intervention, participants will undergo a comprehensive baseline assessment to allow for individualized exercise prescription. The same assessment protocol will be repeated at the end of the 8-week intervention and again at the 4-week follow-up.

The intervention includes:

Eight on-site workshops (one per week during working hours), addressing topics such as musculoskeletal pain management, self-efficacy, physical exercise, mobility, stress management, sleep hygiene, and healthy lifestyle habits.

Two weekly online exercise sessions, delivered asynchronously via a digital platform, focusing on mobility, core stability, and progressive strengthening of the upper and lower limbs and spinal stabilizing muscles.

Exercise programs will be progressive and adapted to participants' perceived exertion and functional capacity. Adherence will be monitored through attendance records and digital tracking of completed exercise sessions. Participants must complete at least 80% of the intervention to be included in the final analysis.

Outcome measures include perceived pain intensity, musculoskeletal symptom prevalence, upper and lower limb muscle strength, physical activity level, work ability, sleep quality, psychosocial factors (stress, anxiety, and depression), health-related quality of life, and work productivity and absenteeism. All measurements are performed using validated instruments and standardized protocols.

ELIGIBILITY:
Inclusion Criteria:

* Have an active employment contract with Lacor Textil covering the entire duration of the study, including the month following the third evaluation phase.
* Be aged 18-65 years (inclusive).
* Be available to participate in all scheduled sessions.

Exclusion Criteria:

* Have severe or specific musculoskeletal conditions that contraindicate exercise.
* Be currently pregnant.
* Be receiving physiotherapy treatment concurrently.
* Be on temporary sick leave during the intervention period.
* Not have the physical capacity required to participate in the workshops and guided exercise.
* Have cognitive or communication impairments that prevent adequate participation.
* Complete less than 80% of the intervention program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity | From baseline to end of treatment (8 weeks) and 4-week follow-up.
  Change in the score on the Numerical Rating Scale (NRS). The NRS scale for pain assessment is a scale that measures the intensity of pain experienced by the patient. It is a numerical rating scale where the patient is asked to rate their pain between 0 and 10. The reported values are classified as follows: no pain = 0; mild pain = 1,2; moderate pain = 3-5; severe pain = 6-8; unbearable pain = 9-10.

SECONDARY OUTCOMES:
Change in Musculoskeletal Symptoms | From baseline to end of treatment (8 weeks) and 4-week follow-up.
  Musculoskeletal disorders will be evaluated using the Standardized Nordic Musculoskeletal Questionnaire (Kuorinka), a self-administered questionnaire consisting of 11 multiple-choice items. The questionnaire provides information on the presence of pain, fatigue, or discomfort in different musculoskeletal body regions. It is designed to detect early musculoskeletal symptoms and to support the analysis of potential ergonomic risk factors. Higher values indicate a greater burden of musculoskeletal symptoms.
Change in Upper Limb Muscle Strength | From baseline to end of treatment (8 weeks) and 4-week follow-up.
  Upper limb muscle strength will be assessed using the handgrip strength test, measured with a hand-held dynamometer (Takei Grip-D). Participants will be seated on a chair with the elbow flexed at 90 degrees and the forearm in a neutral position. Participants will perform a maximal handgrip contraction for up to 3 seconds. Three trials will be conducted, with a 1-minute rest period between attempts. Handgrip strength will be recorded in kilograms (kg), with higher values indicating greater upper limb muscle strength.
Change in Lower Limb Muscle Strength | From baseline to end of treatment (8 weeks) and 4-week follow-up.
  Lower limb muscle strength will be measured using the 30-second Sit-to-Stand-Test (STST).Participants will begin seated on a chair with feet slightly apart and flat on the floor, and arms crossed over the chest. Upon a verbal signal, participants will rise to a full standing position and return to the seated position as many times as possible within 30 seconds. Only correctly completed repetitions, as well as repetitions reaching more than half of the full range of motion at the end of the test, will be counted. Higher numbers of repetitions indicate greater lower limb muscle strength.
Change in Physical Activity Level | From baseline to end of treatment (8 weeks) and 4-week follow-up.
  Physical Activity level will be assessed using the International Physical Activity Questionnaire, Short Form (IPAQ-SF), a validated self-administered questionnaire consisting of 7 items. The questionnaire records the frequency (days per week) and duration (hours and minutes per day) of physical activity performed during a reference week. It is a standardized instrument widely used internationally for population-based physical activity assessment. Higher scores indicate higher levels of physical activity.
Change in Work Ability | From baseline to end of treatment (8 weeks) and 4-week follow-up.
  Work ability will be measured with the Work Ability Index (WAI). The WAI is a self-reporter questionnaire based on the worker's self-perception of their capacity to perform work tasks in relation to job demands and current health status. It includes eleven questions grouped into seven dimensions and generates an overall score reflecting current work ability, as well as an estimation of work ability over the following two years. Higher scores represent better perceived work ability.
Sleep Quality | From baseline to end of treatment (8 weeks) and 4-week follow-up.
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), a 19-item self-administered questionnaire measuring multiple aspects of sleep, including sleep quality, latency, duration, efficiency, disturbances, and daytime dysfunction. Each item is scored to contribute to a global score ranging from 0 to 21, where 0 indicates no sleep difficulties and 21 indicates severe sleep problems. Higher scores reflect poorer sleep quality.
Changes in Depression, Anxiety and Stress | From baseline to end of treatment (8 weeks) and 4-week follow-up.
  Depression, anxiety and stress will be measured with the Depression, Anxiety and Stress Scale (DASS-21). In this scale, each item is answered according to the intensity of each symptom suffered in the last week on a Likert scale from 0 to 3 points. The global scale contains three different blocks for: depression, anxiety and stress. Each block has seven items. The global scale score ranges from 0 to 21 points. In the Depression, Anxiety and Stress Scale, higher scores indicate higher levels of stress, depression and anxiety.
Change in Quality of Life | From baseline to end of treatment (8 weeks) and 4-week follow-up.
  Change in health-related quality of life will be assessed using the EuroQol 5-Dimension 3-Level questionnaire (EQ-5D-3L), Spanish version. The EQ-5D-3L is a validated instrument that can be self-administered or administered via interview to assess health-related quality of life across multiple dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The questionnaire comprises five items, each with three response levels (no problems = 1, some problems = 2, extreme problems = 3). Responses are coded and weighted to generate an index value. Additionally, the EQ-5D-3L includes a 20-centimeter vertical visual analogue scale (VAS) ranging from 0 (worst imaginable health state) to 100 (best imaginable health state), on which participants rate their current perceived health status. Higher scores indicate better health-related quality of life.
Change in Work Absenteeism | From baseline to end of treatment (8 weeks) and 4-week follow-up.
  Work absenteeism will be evaluated using the Work Productivity and Activity Impairment Questionnaire (WPAI), a validated self-administered instrument that measures the impact of health problems on work productivity. The absenteeism domain assesses the percentage of work time missed due to health-related reasons during the previous 7 days. Higher percentages indicate greater work absenteeism.

CONTACTS AND LOCATIONS:
Locations (1):
- Lacor Textil, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers beyond what is included in scientific publications derived from this study. Data sharing is limited to aggregated results presented in peer-reviewed articles to ensure participant confidentiality and comply with data protection regulations.